CLINICAL TRIAL: NCT05099237
Title: A Multi-cohort Trial to Investigate the Feasibility and Acceptability of Wearable Vital Signs Monitors in Patients Undergoing Cancer Treatment in Greater Manchester.
Brief Title: Enhanced Monitoring for Better Recovery and Cancer Experience in Greater Manchester
Acronym: EMBRaCE-GM
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Manchester University NHS Foundation Trust (Other Government)
Collaborators: Zenzium AI Ltd. (Unknown); Aptus Clinical Ltd. (Unknown); The Christie NHS Foundation Trust (Other); University of Manchester (Other); GM Cancer (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Device Feasibility
Other Study IDs: B01227
Record Dates: First submitted 2021-08-26; First posted 2021-10-29 (Actual); Last update posted 2023-05-03 (Actual); Status verified 2023-05

CONDITIONS: Colorectal Cancer; Lung Cancer; Hematological Cancer; CAR T-Cell Therapy
MeSH Terms: conditions — Colorectal Neoplasms; Lung Neoplasms | interventions — Blood Specimen Collection

STUDY DESIGN:
Intervention Model Description: The EMBRaCE-GM study is a multi-cohort trial designed to efficiently evaluate the range of wearable vital signs monitors. Each cohort is a distinct group of patients who undertake a feasibility study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- 1. Colorectal Cancer (Active Comparator): This cohort seeks to investigate the feasibility of using two commercially available health and wellbeing trackers to monitor patients with colorectal cancer who are about to start treatment. Participants will be asked to:
  * Wear the OURA ring and the Withings ScanWatch for the duration of their planned cancer treatment up to a maximum of 26 weeks (6 months).
  * Complete weekly wearable device satisfaction surveys and weekly cancer specific patient reported outcomes measures (modified FACT-C survey).
  * Report specific symptoms on an ad-hoc basis as they wish.
  Interventions: Device: OURA Ring; Device: WithingsScan Watch; Other: Quality of Life Surveys
- 2. Lung Cancer (Active Comparator): This cohort seeks to investigate the feasibility of using two commercially available health and wellbeing trackers to monitor patients with lung cancer who are about to start treatment. Participants will be asked to:
  * Wear the OURA ring and the Withings ScanWatch for the duration of their planned cancer treatment up to a maximum of 26 weeks (6 months).
  * Complete weekly wearable device satisfaction surveys and weekly cancer specific patient reported outcomes measures (modified FACT-L survey).
  * Report specific symptoms on an ad-hoc basis as they wish.
  Interventions: Device: OURA Ring; Device: WithingsScan Watch; Other: Quality of Life Surveys
- 3. Haematological Cancer (Active Comparator): Participants (with haematological malignancy about to start treatment with CAR T-cell therapy or another cellular therapy product) will be asked to:
  * Wear an OURA ring and Withings ScanWatch for approx five weeks including whilst they are in hospital (prior to CAR T-cell therapy and continue for 28 days post infusion)
  * Wear an Isansys LifeTouch, Isansys LifeTemp and Nonin Model 3150 WristOx™ Pulse Oximeter during their inpatient stay only, up to a maximum of 28 days.
  * Supported to take daily weights using Withings Body Scale.
  * Asked to complete weekly electronic quality of life surveys
  * Provide a series of 12 blood samples to measure inflammatory molecules at various intervals
  Interventions: Device: OURA Ring; Device: WithingsScan Watch; Drug: Isansys Patient Status Engine; Other: Quality of Life Surveys; Diagnostic Test: Blood Samples; Other: Daily Weights

INTERVENTIONS:
Device: OURA Ring — All participants will be asked to wear an OURA ring and WithingsScan Watch both at home and whilst in hospital. These devices can record activity, sleep type and duration, resting heart rate and heart rate variability along with a range of other vital signs.
Device: WithingsScan Watch — All participants will be asked to wear an OURA ring and WithingsScan Watch both at home and whilst in hospital. These devices can record activity, sleep type and duration, resting heart rate and heart rate variability along with a range of other vital signs.
Drug: Isansys Patient Status Engine — Participants in cohort 3 will also be asked to wear Isansys monitoring devices whilst they are in hospital. They will begin to wear the monitors prior to CAR T-cell therapy and continue for 28 days post infusion. Participants will be asked to wear an Isansys LifeTouch, Isansys LifeTemp and Nonin Model 3150 WristOx™ Pulse Oximeter during their inpatient stay only, up to a maximum of 28 days.
  Arms: 3. Haematological Cancer
Other: Quality of Life Surveys — On a weekly basis participants will be asked to complete satisfaction surveys for the devices they are wearing (ring and watch) and report on their quality of life through standardised questionnaires. These surveys will be delivered electronically to participants via their smartphone or tablet device. There will be an option for participants to report adhoc symptoms via an app on their smartphone or tablet device.
Diagnostic Test: Blood Samples — COHORT 3 ONLY
  Participants in Cohort 3 only will be asked to provide a series of blood samples to measure inflammatory molecules during the study. These will be requested at various intervals during face-to-face visits and whilst the patient is in hospital:
  * Baseline blood sample during study enrolment
  * Post-lymphodepletion and prior to CAR T-cell infusion (this may be on day -1 or day 0 as needed)
  * Post CAR T-cell infusion:
    * Day 1
    * Day 3
    * Day 6
    * Day 9
    * Day 14 (if the participant remains in hospital)
  A sample of blood will be taken at baseline and a further sample post lymphodepletion and prior to CAR T-cell infusion. Post CAR T-cell infusion, samples will be taken at two timepoints (morning and afternoon) on each of the sampling days.
  Arms: 3. Haematological Cancer
Other: Daily Weights — COHORT 3 ONLY
  During their inpatient stay, up to a maximum of 28 days, participants in Cohort 3 will be supported to weigh themselves daily using a Withings Body Scale.
  Arms: 3. Haematological Cancer

SUMMARY:
The EMBRaCE-GM study is a multi-cohort trial designed to efficiently evaluate the range of wearable vital signs monitors that could be used to support patients during cancer treatment.

The aims of the study are to determine

* to determine if continuous vital signs monitoring is feasible during cancer treatment
* to determine if such monitoring is acceptable to patients undergoing cancer treatment
* to determine what insights could be made with the data obtained

A multi-cohort study is essential because there are a huge range of vital signs monitors that could be useful and a method that allows quickly identification of the devices that are most acceptable to patients and which offer the most useful information to clinicians is needed. Similarly, the best device may vary according to the specific disease and the treatment a patient is offered.

Each cohort in the study will investigate a variety of wearable vital signs monitors in different patient groups undergoing different treatments. A common data collection platform will be used for all cohorts with a modular design that allows data collection to be adapted slightly to meet specific needs for each cohort.

DETAILED DESCRIPTION:
1 in 2 people will be diagnosed with cancer during their lifetime with over 350,000 new cancer diagnoses per year (UK). Cancer treatment is a complex process. Patients experience a range of symptoms as a consequence of their disease and their treatment. Sometimes, the treatment itself can lead to specific life-threatening complications.Patients who recover may be left with lasting physical and psychological consequences. A third of those who are suffering from cancer or who have recovered from it classify their health as 'average to poor' which is double the rate reported by individuals without health problems. There is an ongoing need to offer patients personalised support through their cancer journey and to identify and minimise complications.

This need for personalised cancer care is emphasised in the NHS Long Term Plan (2019). A key aim of which is to improve cancer survival but with a focus on giving patients 'more control over their health' through improved self-management. The long-term plan identifies a need for digitally-enabled care to empower patients and highlights that artificial intelligence (AI) and digital clinical decision support could play a role in this regard.

Wearable vital signs monitors offer a solution by which patients can be monitored more frequently and in more detail during cancer treatment. There is a huge variety of wearable monitors which range from commercially available well-being trackers to CE marked medical devices. The devices themselves take many forms which may vary in their acceptability to patients and utility to health care professionals. The parameters which can be monitored range from traditional vital signs to more holistic measures of sleep, stress and activity. Such information could help to identify individuals who are recovering well, those who are experiencing specific symptoms or those who need extra assistance.

The availability of commercial well-being monitors is growing rapidly and monitors are becoming progressively more sophisticated. Monitors are also increasingly used in medical research in conjunction with or in place of formal medical devices. This trend has been highlighted in a recent systematic review in which the authors noted the need for further research to understand the validity and acceptability of using such devices in an outpatient healthcare setting. This is particularly true for patients suffering from cancer, where the vast majority of wearable device research has focused upon exercise trackers, the breast cancer tumour type and patients who have already completed their cancer treatment. In addition, the acceptability of such devices to patients has been shown to vary. The COMPARE study reported that patients are broadly supportive of artificial intelligence (AI) and wearable devices whilst a study in patient genitourinary cancer found that acceptability of wearable devices varied between 100% (40-49 years) and 40% (80-89 years).

The situation is broadly the same for wearable vital signs monitors which are registered as medical devices. Whilst these devices have been more extensively studied, the majority of research does not pertain to cancer patients and no specific use case has been identified in this patient population.

Therefore, before wearable vital signs monitors can play a role in cancer care it is essential that the acceptability of the range of devices is formally evaluated in a variety of cancer types, in a broad demographic of patients, over the duration of cancer treatment and in a variety of treatment modalities and settings. The investigators aim to understand the potential of these devices to offer new insights and learn if the information provided can be useful to patients and healthcare professionals.

ELIGIBILITY:
Inclusion Criteria:

All individuals who participate in the EMBRaCE-GM study will have capacity to consent to enrol in the study at the point of screening and consent. This is an inclusion criteria for the study.

Cohort 1 -

Individuals are eligible to be included in the study only if all the following criteria apply:

* Adult (aged 16 years or older)
* Diagnosis of colorectal cancer confirmed at MDT
* Active treatment planned which must include surgery
* The individual is aware of the confirmed diagnosis and understands the proposed treatment plan.
* Owns a smart phone/tablet compatible with the OURA ring and Withings ScanWatch and is willing to have the OURA app and Withings app installed on their device.
* The patient has an email account or is willing to create one to register with the OURA and Withings apps.
* Capable of charging and managing the wearable sensors (OURA ring and Withings ScanWatch) at home

Cohort 2 -

Individuals are eligible to be included in the study only if all of the following criteria apply:

* Adult (aged 16 years or older)
* Diagnosis of lung cancer confirmed at MDT
* Active treatment planned
* The individual is aware of the confirmed diagnosis and understands the proposed treatment plan.
* Owns a smart phone/tablet compatible with the OURA ring and Withings ScanWatch and is willing to have the OURA app and Withings app installed on their device.
* The patient has an email account or is willing to create one to register with the OURA and Withings apps.
* Capable of charging and managing the wearable sensors (OURA ring and Withings ScanWatch) at home

Cohort 3 -

Individuals are eligible to be included in the study only if all the following criteria apply:

Adult (aged 16 years or older)

* Consented to receive a CAR T-cell therapy or other cellular therapy product for treatment of a haematological malignancy.
* The individual is aware of the confirmed diagnosis and understands the proposed treatment plan.
* Owns a smart phone/tablet compatible with the OURA ring and Withings ScanWatch/Smart Scale and is willing to have the OURA app and Withings app installed on their device.
* The patient has an email account or is willing to create one to register with the OURA and Withings apps.
* Capable of charging and managing the wearable sensors (OURA ring and Withings ScanWatch) at home

Exclusion Criteria:

Cohort 1 & Cohort 2 -

Individuals are excluded from the study if any of the following criteria apply:

* Patients unable to give informed consent.
* Patients in whom treatment is limited to "best supportive care"
* Patients with cognitive or sensory deficits that would prevent them from following instructions and using the wearable device correctly/as instructed.
* Patients for whom there is no suitably sized OURA ring or Withings ScanWatch available at the time of screening*.
* Patients who are non-English speakers - an essential requirement to interact with the wearable device apps and complete the web-based surveys that form part of the study.

Cohort 3 -

Individuals are excluded from the study if any of the following criteria apply:

* Patients unable to give informed consent.
* Patients in whom treatment is limited to "best supportive care"
* Known allergy or history of contact dermatitis to medical adhesives.
* Patients with pacemakers, implantable defibrillators or neurostimulators.
* Patients with prion related diseases e.g., Spongiform Encephalopathies
* Patients with cognitive or sensory deficits that would prevent them from following instructions and using the wearable device correctly/as instructed.
* Patients for whom there is no suitably sized OURA ring or Withings ScanWatch available at the time of screening*.
* Patients who are non-English speakers - an essential requirement to interact with the wearable device apps and complete the web-based surveys that form part of the study.

For all cohorts -

* It is essential that participants wear appropriately sized OURA rings and Withings ScanWatches to ensure that they are comfortable and that the data collected is accurate. The study has purchased enough rings and watches to ensure that the majority of participants can be easily accommodated but on rare occasions a suitably sized device may not be available.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2021-12-01 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Cohort 1/2 - Primary outcome measure: feasibility of monitoring for each wearable monitor (ring and watch): | Maximum of 6 months
  The proportion of participants who completed the planned duration of monitoring with the device (ie:- did not request to terminate the study early) and the amount of time vital signs were actually recorded by the device expressed as a percentage of the total time the patient wore the device on the study.
Cohort 3 - Primary outcome measure: feasibility of monitoring for the OURA ring and Withings ScanWatch: | 5 weeks
  The proportion of participants who completed 5 weeks of monitoring and the full period of monitoring (hospital admission to discharge, max 28 days) with the device (i.e:- did not request to remove the device early) as the amount of time vital signs were actually recorded by the device expressed as a percentage of the total duration of the participant's planned cancer treatment.
Cohort 3 - Primary outcome measure: feasibility of monitoring for the Isansys medical devices LifeTouch, LifeTemp and Nonin Pulse Oximeter): | Maximum of 28 days
  The proportion of participants who completed 5 weeks of monitoring and the full period of monitoring (hospital admission to discharge, max 28 days) with the device (i.e:- did not request to remove the device early) as the amount of time vital signs were actually recorded by the device expressed as a percentage of the total time the patient wore the device on the study.
Cohort 3 - Primary outcome measure: feasibility of monitoring for the daily weights: | Maximum of 28 days
  The number of daily weights recorded (inpatient stay, max 28 days)

SECONDARY OUTCOMES:
Cohorts 1,2 and 3 Device acceptability | through study completion, an average of 6 months
  The outcome is measured as an overall device acceptability to participants, this will be reflected as the number of eligible patients who declined to take part in the study and their reasons for declining compared to participant feedback of acceptability.
Cohorts 1,2 and 3 Device acceptability | through study completion, an average of 6 months
  Participants will be asked to complete a weekly survey (via smart phone/tablet) to determine the acceptability of the devices to patients:
  - Likert scale acceptability ratings for each wearable monitor(pre-defined answer options, ranging from "very likely" through to "highly unlikely" on a 5-point scale) and free text comments on wearing the devices
Cohorts 1,2 and 3 Device acceptability | through study completion, an average of 6 months
  Participants will be asked to complete a weekly survey (via smart phone/tablet) to determine the acceptability of the devices to patients:
  - The percentage of participants who report each week that they have decided to stop wearing the device (via weekly survey) and categorical reasons for device removal (via weekly survey)
Cohorts 1,2 and 3 Device acceptability | through study completion, an average of 6 months
  Participants will be asked to complete a weekly survey (via smart phone/tablet) to determine the acceptability of the devices to patients:
  - The percentage of the devices that are successfully returned for re-use at the end of the study period and for devices that were not returned, what was the reason for this?
Cohorts 1,2 and 3 Device acceptability | through study completion, an average of 6 months
  Participants will be asked to complete a weekly survey (via smart phone/tablet) to determine the acceptability of the devices to patients:
  - Likert scale ratings (pre-defined answer options, ranging from "very likely" through to "highly unlikely" on a 5-point scale) and free text comments concerning the extent to which the devices support self-management.

CONTACTS AND LOCATIONS:
Overall Officials: Dr Anthony Wilson, Principal Investigator — Manchester University NHS Foundation Trust
Locations (1):
- Manchester University NHS Foundation Trust, Manchester, United Kingdom

IPD SHARING:
Plan to Share IPD: No